CLINICAL TRIAL: NCT01361256
Title: Pilot Study of WA-NG Telescope Prosthesis in Patients With Central Vision Impairment Associated With End-stage Age-related Macular Degeneration
Brief Title: Study of WA-NG Telescope Prosthesis in Patients With End-stage Age-related Macular Degeneration
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA-NG-001
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2016-10

CONDITIONS: Age Related Macular Degeneration
Keywords: Macular Degeneration; Visual Impairment; Implantable Telescope
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WA- NG Telescope Prothesis (Experimental): Implantable Miniature Telescope for end stage AMD (Age-related Macular Degeneration)
  Interventions: Device: Telescope prosthesis; Device: WA-NG Telescope Prothesis

INTERVENTIONS:
Device: Telescope prosthesis — Monocular implantation of the telescope prosthesis after cataract extraction
  Other Names: IMT-NG
Device: WA-NG Telescope Prothesis — The WA-NG telescope prosthesis (Figure 1) is the next generation telescopic implantable device which, when combined with the optics of the cornea, constitutes a telephoto system for improvement of visual acuity in patients with severe to profound vision impairment due to bilateral, end-stage age-related macular degeneration. The device is implanted in one of the patient's eyes. In this way, the implanted eye provides central vision and the non-implanted eye can continue to provide peripheral vision.

SUMMARY:
This is a pilot study to evaluate the safety of the Model WA-NG telescope prosthesis in patients with bilateral moderate to profound central vision impairment due to end-stage age-related macular degeneration.

DETAILED DESCRIPTION:
Patients will be screened for eligibility and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible patients will be examined preoperatively to obtain a medical history and to establish a baseline for ocular condition. Baseline measurements will include successful use of an external telescope.

Postoperatively, patients will undergo ophthalmic evaluation at regular intervals as specified in this protocol and will be required to return for 6 to 10 additional visits for vision training with a low vision specialist.

ELIGIBILITY:
Inclusion Criteria:

* Bi-lateral, stable, moderate to profound (20/80 to 20/800) central vision impairment due to bilateral scotoma associated with end-stage macular degeneration, defined as retinal finds of bilateral, geographic atrophy or disciform scar with foveal involvement. Phakic in the operative eye. Must achieve a 5 letter improved with external telescope simulator. More medical

Exclusion Criteria:

* Evidence of active CNV or any ophthalmic pathology that compromises peripheral vision of fellow eye or predisposes eye rubbing. Previous intraocular of corneal surgery of any kind in operative eye. Retinal disease, optic nerve disease, diabetic retinopathy, retinal tears, or any intraocular tumor or medical or ophthalmic condition that in the opinion of the investigator renders the subject unsuitable for participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Positional Stability | 12 months
  Positional stability assessed by slit lamp examination and anterior segment OCT

SECONDARY OUTCOMES:
Adverse events | 12 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mordecai Rosner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Hasomer, Israel